CLINICAL TRIAL: NCT04778111
Title: Segmental Exclusion of the Upper Limb and Peri-personal Space
Acronym: EPPEX
Status: Completed | Type: Observational
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Other Study IDs: IRR-CLP-2021-3
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Patients With Musculoskeletal Disorders of the Upper Limb With Symptoms of Exclusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with exclusion
  Interventions: Other: Measurement of the actual and perceived maximum reachable distance
- Control
  Interventions: Other: Measurement of the actual and perceived maximum reachable distance

INTERVENTIONS:
Other: Measurement of the actual and perceived maximum reachable distance — A device (a table) will present luminous targets (green circles) to the subjects. Subjects will be asked to determine whether or not they are able to reach this target with their upper limb.

SUMMARY:
This study is based on previous studies on the search of the limit of the peri-personal space. In a previous study, Gouzien et al. (2017) evaluated the peri-personal space of action of patients with upper limb amputations and sought a link between this space and the level of integration of their myoelectric prosthesis. We have decided to implement part of this protocol to evaluate the peri-personal space for another population with upper limb patholog: segmental exclusion of the upper limb.

Exclusion is a phenomenon that is very little studied but known to orthopedic surgeons and physical medicine and rehabilitation physicians. It is characterized by the non-use or underuse of a limb segment in the absence of central nervous system involvement. This phenomenon is compared to peripheral neglect. Most of the time, the patient is unaware of his disorder "he forgets his finger without realizing it", but this phenomenon can be reversible under verbal exhortation from a third party.

The aim of this study is to observe if there is a change in peri-personal space in patients with unilateral segmental exclusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age greater than or equal to 18 years old).
* Person with a symptom of unilateral exclusion.
* Person with no contraindication to hard work in activities of daily living due to the lesions.
* Person who has given informed consent.

Exclusion Criteria:

* Person under 18 years of age.
* Person with visual impairment
* A person with a central neurological pathology.
* A person with cognitive impairment related to a brain injury, psychiatric illness or intellectual disability.
* A person who has difficulty understanding instructions.
* A person of full age who is subject to a legal protection measure or who is unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients included in this study are patients with upper extremity musculoskeletal disorders of traumatic origin. To these disorders is added a segmental exclusion syndrome, which is defined as the under-use or non-use of part of the upper limb.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Delta-MRD | During one evaluation session
  Difference (in cm or in % of error) between actual maximum reachable distance and perceived maximum reachable distance

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France

IPD SHARING:
Plan to Share IPD: No